CLINICAL TRIAL: NCT00188760
Title: Optical Quantification of Breast Density Changes Due to Hormone Treatment, Pregnancy and Breast-feeding.
Brief Title: Breast Study Investigating a New Light Technique to Monitor Changes in Breast Tissue Density
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: Susan G. Komen Breast Cancer Foundation (Other); Dr. Julia Knight (research collaborator) (Unknown)
Responsible Party: Dr. Lothar Lilge, University Health Network
Other Study IDs: UHNREB#02-0712-C; SGKBCF#BCTR0402530; MSHREB#02-0226-E; UTREB#9313; HC#69745
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2011-10-07 (Estimated); Status verified 2011-10

CONDITIONS: Breast Cancer
Keywords: Breast Transillumination Spectroscopy; Optical Transillumination Spectroscopy; Breast Cancer Risk
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to test the ability of a technique called Transillumination Breast Spectroscopy (TIBS) to monitor an individual's breast density changes over time.

DETAILED DESCRIPTION:
Breast density is an established physical risk factor for breast cancer, applicable to the entire female population in a pre-breast-screening program and, unlike other risk factors, was shown to be affected by an intervention treatment. High breast tissue density is associated with increased risk of breast cancer. Transillumination Breast Spectroscopy (TIBS) uses a white light to provide spectral information on breast tissue density and composition (e.g. water, lipid, hemoglobin and other biomolecules). The overall goal of the TIBS program is to develop a technique that can identify individuals at high risk for breast cancer who would benefit most from improved screening methods and a risk reducing intervention (e.g. diet and lifestyle changes) and can monitor the efficacy of the risk reducing intervention itself in an individual. In a previous study, we demonstrated a high correlation between breast density assessed by TIBS and density identified by x-ray mammography. The current study is testing TIBS ability to monitor changes in an individual's breast density over time

ELIGIBILITY:
Inclusion Criteria:

* Be in good health and able to provide consent
* Be between 25 and 45 years of age
* Be pre-menopausal
* Are willing to come in to Princess Margaret Hospital (Toronto, Ontario, Canada) for up to 12 visits at intervals of about three months

Exclusion Criteria:

* Have had a full term pregnancy
* Have had breast biopsy
* Have had breast augmentation or reduction

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Cases recruited from the Reproductive Biology Unit at Mount Sinai Hospital and the University Health Network community. Controls recruited from University Health Network community and the University of Toronto community. (Toronto, Ontario, Canada)
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2004-05; Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lothar Lilge, PhD, Principal Investigator — Ontario Cancer Institute, University Health Network, Toronto, Ontario, Canada M5G 2M9; Department of Biophysics and Bioimaging, University of Toronto, Ontario, Canada M5G 2M9
Locations (1):
- Ontario Cancer Institute, Princess Margaret Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Blyschak K, Simick M, Jong R, Lilge L. Classification of breast tissue density by optical transillumination spectroscopy: optical and physiological effects governing predictive value. Med Phys. 2004 Jun;31(6):1398-414. doi: 10.1118/1.1738191. PMID 15259643
- [Background] Simick MK, Jong R, Wilson B, Lilge L. Non-ionizing near-infrared radiation transillumination spectroscopy for breast tissue density and assessment of breast cancer risk. J Biomed Opt. 2004 Jul-Aug;9(4):794-803. doi: 10.1117/1.1758269. PMID 15250768
- [Background] Blackmore KM, Knight JA, Jong R, Lilge L. Assessing breast tissue density by transillumination breast spectroscopy (TIBS): an intermediate indicator of cancer risk. Br J Radiol. 2007 Jul;80(955):545-56. doi: 10.1259/bjr/26858614. Epub 2007 May 30. PMID 17537757
- [Background] Simick MK, Lilge L. Optical transillumination spectroscopy to quantify parenchymal tissue density: an indicator for breast cancer risk. Br J Radiol. 2005 Nov;78(935):1009-17. doi: 10.1259/bjr/14696165. PMID 16249602